CLINICAL TRIAL: NCT03005509
Title: Structured Trauma Quality Improvement Meetings at Four Trauma Centres in India: Protocol for a Prospective Observational Study to Assess Effectiveness
Brief Title: Structured Trauma Quality Improvement Meetings at Four Trauma Centres in India
Acronym: TQI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr Gerard O'Reilly (Other)
Collaborators: National Trauma Research Institute (Other); The Alfred (Other); Monash University (Other); All India Institute of Medical Sciences (Other); The George Institute for Global Health, Australia (Other); Sheth Vadilal Sarabhai General Hospital (Other); Guru Teg Bahadur Hospital (Other); Lokmanya Tilak Municipal Medical College and Hospital (Other); Centralised Accident and Trauma Services, Delhi, India (Other Government); GVK EMRI: Emergency Management and Research Institute (Other); Maharashtra Emergency Medical Services, India (Other); Nathiba Hargovandas Lakhmichand Municipal Medical College, India (Unknown); University College of Medical Sciences, India (Individual)
Responsible Party: Sponsor-Investigator, Dr Gerard O'Reilly, Principal Investigator, National Trauma Research Institute
Organization: National Trauma Research Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GCF020013-TQI
Record Dates: First submitted 2016-12-19; First posted 2016-12-29 (Estimated); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Major Trauma; Injuries Major
Keywords: Quality improvement; Injury; Injuries
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-intervention group (No Intervention): All injured patients to the four intervention sites) and allocated to a red (1st) or yellow (2nd) priority triage category will be eligible for inclusion.
  The Trauma Quality Improvement Meeting (TQIM) checklist will not be introduced during this phase.
- Post-intervention group (Other): All injured patients to the four intervention sites) and allocated to a red (1st) or yellow (2nd) priority triage category will be eligible for inclusion.
  The Trauma Quality Improvement Meeting (TQIM) checklist will be used at all Trauma Quality Improvement Meetings (TQIMs)
  Interventions: Other: TQIM checklist

INTERVENTIONS:
Other: TQIM checklist — The intervention phase will include an intense training period covering:
  1. Conduct of Trauma Quality Improvement Meeting (TQIM) (and Trauma Quality Improvement program in general). The training will be delivered using the World Health Organization (WHO) Trauma Quality Improvement Programmes short course and online resources.
  2. Implementation of Trauma Quality Improvement Meeting (TQIM) Checklist.
  Other Names: Structured TQI program
  Arms: Post-intervention group

SUMMARY:
A prospective before-and-after study to evaluate the effect of implementing a Trauma Quality Improvement protocol on the process of Trauma Quality Improvement meetings and major trauma patient outcomes at four trauma centres in India.

DETAILED DESCRIPTION:
This project will be conducted as a prospective before-and-after study at four major trauma centres in India, with the intervention occurring between pre- and post-intervention phases. Included in the study will be all patients presenting to any of the four trauma hospitals with a potentially life-threatening or limb-threatening injury. The intervention will be the introduction of a structured Trauma Quality Improvement Meeting (TQIM), using a checklist and training program. The primary outcome will be compliance with the TQIM checklist, measured as the proportion of discussed cases (trauma deaths) for which problems with care, preventability and corrective actions were discussed and / or agreed. The secondary outcomes will include in-hospital risk-adjusted mortality, hospital length of stay and time to emergency surgery. Data collection will occur at all meetings at the four trauma hospitals at which trauma deaths are discussed. Data will also be collected in a dedicated trauma registry.

ELIGIBILITY:
Inclusion Criteria:

* All patients presenting to any of the four study sites with a potentially life-threatening or limb-threatening injury. Specifically, all presenting injured patients triaged as "Red" or "Yellow" according to the Australia-India Trauma Systems Collaboration (AITSC) Trauma Triage Protocol, will meet the screening criteria for data collection. Retrospective inclusion in the registry will be continued for all screened patients presenting to any of the included hospitals with injury (including near-drowning) as the primary diagnosis and with at least one of the following criteria:

  * Admission to hospital
  * Death after triage but before admission

Exclusion Criteria:

* The exclusion criteria for the AITSC Trauma Registry are:

  * Death at scene
  * Alive at triage but not admitted to hospital
  * Isolated poisoning
  * Isolated burns
  * Single digit finger or toe amputations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2017-01; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
TQIM Checklist compliance - preventability | Up to 14 months
  TQIM Checklist compliance - % of cases for which it is agreed that care can be improved

SECONDARY OUTCOMES:
TQIM Checklist compliance - corrective action | Up to 14 months
  TQIM Checklist compliance - % of cases (where it is agreed that care can be improved) for which at least one corrective action is agreed
In hospital risk-adjusted mortality | Up to 14 months
  In-hospital risk-adjusted mortality: The proportion of deaths amongst those with Injury Severity Score (ISS) >12 and <50.
Hospital length of stay | Up to 14 months
  Hospital length of stay
Time to emergency surgery | Up to 14 months
  Time from hospital arrival to operating theatre for patients undergoing emergency surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Fitzgerald, MBBS, MD, Principal Investigator — National Trauma Research Institute
Locations (4):
- India (4):
  - Vadilal Sarabhai Hospital, Ahmedabad, Gujarat
  - Lokmanya Tilak Municipal General Hospital, Mumbai
  - Guru Teg Bahadur Hospital, New Delhi
  - JPN Apex Trauma Centre at All India Institute of Medical Sciences, New Delhi

IPD SHARING:
Plan to Share IPD: No